CLINICAL TRIAL: NCT04160624
Title: The Effect of Transcatheter Aortic Valve Replacement With Extracorporeal Life System Support to Cure Aortic Stenosis/Regurgitation Patients
Brief Title: Transcatheter Aortic Valve Replacement With Extracorporeal Life System Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Jian Yang, Deputy chief surgeon, Xijing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xjyyxwk002
Record Dates: First submitted 2019-11-01; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Aortic Stenosis; Aortic Regurgitation; Heart Failure With Reduced Ejection Fraction
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement; Extracorporeal Membrane Oxygenation; Cardiopulmonary Bypass

STUDY DESIGN:
Intervention Model Description: ECLS-assisted TAVR for patients with very low EF(<20%). Only TAVR for patients with fair EF(>20%)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-ECLS GROUP (Active Comparator): For AS/R patients with normal EF, only TAVR was performed
  Interventions: Procedure: transcatheter aortic valve replacement
- ECLS GROUP (Experimental): For AS/R patients with low EF, TAVR under ECLS-assisted was performed
  Interventions: Procedure: transcatheter aortic valve replacement

INTERVENTIONS:
Procedure: transcatheter aortic valve replacement — Use Venus-A valve or J-Valve to perform TAVR procedure. Use cardiopulmonary bypass or cardiopulmonary bypass to provide ECLS
  Other Names: extracorporeal life support system; extracorporeal membrane oxygenation; cardiopulmonary bypass

SUMMARY:
Transcatheter aortic valve replacement (TAVR) has a high risk and a high mortality rate in the treatment of aortic stenosis/regurgitation patients with cardiac insufficiency. The investigators aim to discuss the clinical efficacy of extracorporeal life support system(ECLS) during TAVR procedure in severe aortic lesion under very low ejection fraction (EF).

DETAILED DESCRIPTION:
Transcatheter aortic valve replacement (TAVR), characterized by minimal invasion, no need for thoracotomy and extracorporeal circulation and definite mid- and long-term efficacy, has been recognized as an effective alternative replacing valve replacement through conventional thoracotomy for senile aortic valve stenosis. However, there are still a large number of patients whose left ventricular ejection fraction (LVEF) significantly declines due to the long history of disease and long-term heart injury, entering the decompensation stage. TAVR will still lead to such severe complications as intraoperative hemodynamic collapse and malignant arrhythmia in these patients, greatly increasing the mortality rate. It is pointed out in the American Heart Association Guideline (2017) that TAVR is not recommended as a treatment means for patients with very poor cardiac function under EF <20%. After conservative medication, the prognosis of patients with aortic valve stenosis under very low EF is poor with a 3-year mortality rate above 85%, and the prognosis after heart transplantation remains controversial. According to the pathological basis of patients and preoperative results of dobutamine test, the cardiac systolic function of some patients is expected to be significantly improved after removal of aortic valve stenosis. Therefore, applying extracorporeal life support system, such as extracorporeal membrane oxygenation (ECMO) or cardiopulmonary bypass (CPB） in the guarantee of cardiopulmonary function during perioperative period of TAVR is considered as the optimal surgical strategy for such patients.

ELIGIBILITY:
Inclusion Criteria:

1. The age of patient is ≥50 yrs;
2. Severe aortic stenosis or regurgitation patients (The area of central regurgitation exceeds 40% of left ventricular area; regurgitant volume ≥10ml；EROA≤1.0cm2; PGmean≥50mmHg (Satisfy any condition).
3. Small incision surgery of chest can be tolerated.
4. General anesthesia is tolerable

4. The subject was informed of the clinical application nature of the technology and agreed to participate in all requirements of the clinical application of the new technology, signed the informed consent and agreed to complete.

Exclusion Criteria:

1. Subject who are pregnant, lactating or scheduled to pregnant during the period of the clinical new technology.
2. Subjects with active endocarditis or rheumatic mitral valve disease.
3. Life expectancy <1 year for cardiac or other malignant tumors.
4. Participate in other clinical trial.
5. In the judgment of the investigator, subjects had poor acceptance of chemotherapy, and they cannot complete the trial as required.

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiac event | 1 year
  Include by limited to: death, emergency surgery, surgically related stroke, severe bleeding, rehospitalization, redo surgery

SECONDARY OUTCOMES:
minor adverse event | 1 year
  Include by limited to: perivalvular regurgitation, infection, arrhythmia, Peripheral vascular complications

CONTACTS AND LOCATIONS:
Overall Officials: Shiqiang Yu, M.D. PH.D., Principal Investigator — The First Affiliated Hospital of Air Force Medicial University
Locations (1):
- Department of Cardiovascular Surgery of Xijing Hospital, Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No